CLINICAL TRIAL: NCT03389451
Title: 68Ga PSMA-HBED-CC PET in Patients With Biochemical Recurrence
Brief Title: 68Ga PSMA PET for Patients With Biochemical Recurrence of Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michael Graham PhD, MD (Other)
Collaborators: University of Iowa (Other); Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Michael Graham PhD, MD, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201709730
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Prostatic Neoplasm; Prostatic Neoplasms, Castration-Resistant; Prostatic Cancer Recurrent; Prostatic Cancer Metastatic
Keywords: 68Ga-PSMA-11; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga PSMA-HBED-CC
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga PSMA PET scan (Experimental): Ga-68 PSMA-HBED-CC PET
  Interventions: Drug: Ga-68 PSMA-HBED-CC PET

INTERVENTIONS:
Drug: Ga-68 PSMA-HBED-CC PET — Ga-68 PSMA-HBED-CC is an investigational PET drug (radionuclide), that binds to the prostate specific receptors. The dose will be about 5mCi (range 3-7 mCi) and administered intravenously.
  Other Names: Gallium-68 PSMA-HBED-CC PET scan

SUMMARY:
This study investigates if a new prostate-specific membrane antigen (PSMA) drug makes prostate cancer easier to identify in positron-emission tomography (PET) imaging. If this works, prostate cancer treatments can be prescribed that match the location of the disease. PSMA is radiolabeled with Gallium-68 (Ga-68). This means a participant receives a small dose of radiation from the drug - less than the annual radiation limit for a medical worker.

To test this new drug, participants will receive an injection of Ga-68 PSMA and then have a PET scan. This PET scan, and the reported results, will be entered into the medical record and shared with the treating oncologists.

DETAILED DESCRIPTION:
This study evaluates PSMA-HBED-CC labelled with Gallium-68, abbreviated 68Ga PSMA. This is a radiotracer that attaches to receptors in the membrane of prostate cancer cells. The 68Ga PSMA is identified using a positron emission tomography (PET) scanner. It is believed that 68Ga PSMA will identify prostate cancer more precisely than normal imaging methods (MRI, CT, or ultrasound). Imaging is key to successful treatment - disease must be identified to be treated.

Men who have biochemical recurrence of prostate cancer are invited to test 68Ga PSMA. Participants undergo the 68Ga PSMA PET scan before further treatment. Clinical information, including any MRI, CT, or ultrasound imaging and biopsy/surgery information, will be used to determine if the 68Ga PSMA PET imaging was better than the standard imaging. The study team will collect this information for about 1 year after the PSMA scan.

Depending on findings, participants may be invited back for a second 68Ga PSMA scan. This is done if the first scan showed positive lymph nodes or soft tissue metastases but a surgery or biopsy result does not.

The results from these scans will be shared with the participant. Results will also be entered into the participant's medical record and shared with the treating oncologists.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven prostate adenocarcinoma
* Rising prostate-specific antigen (PSA )after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy)
* If post-radical prostatectomy, PSA > 0.2 ng/mL measured > 6 weeks post-operative and confirmed persistent PSA > 0.2 ng/mL (AUA recommendation for biochemical recurrence)
* If post-radiation therapy, PSA that is ≥ 2 mg/mL rise above PSA nadir (ASTRO recommendation for biochemical recurrence)
* Not receiving any other investigational agents (i.e., unlabeled drugs or drugs under an IND for initial efficacy investigations)
* No other malignancy within the past 2 years (skin basal cell or cutaneous superficial squamous cell carcinoma or superficial bladder cancer are exempt from this criterion)
* Karnofsky performance status (KPS) ≥ 50 (ECOG/WHO of 0, 1, or 2)
* Ability to understand and willingness to provide informed consent

Exclusion Criteria:

* Cannot receive furosemide
* History of Stevens Johnson syndrome
* History or diagnosis of Paget's disease
* Malignancy other than current disease under study
* Allergy to sulfa or sulfa-containing medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Graham, MD, PhD, Study Chair — University of Iowa
Locations (1):
- The University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Codified data will be archived and stored in an imaging repository with limited metadata for analysis. Individuals seeking use of these data should contact the study chair. A data sharing contract for a HIPAA limited dataset will need to be executed prior to data sharing.
Supporting Information: CSR
Time Frame: Available as requested. Data will be archived indefinitely for research purposes.
Access Criteria: Individuals seeking use of these data should contact the study chair.

REFERENCES:
- [Background] Maurer T, Gschwend JE, Rauscher I, Souvatzoglou M, Haller B, Weirich G, Wester HJ, Heck M, Kubler H, Beer AJ, Schwaiger M, Eiber M. Diagnostic Efficacy of (68)Gallium-PSMA Positron Emission Tomography Compared to Conventional Imaging for Lymph Node Staging of 130 Consecutive Patients with Intermediate to High Risk Prostate Cancer. J Urol. 2016 May;195(5):1436-1443. doi: 10.1016/j.juro.2015.12.025. Epub 2015 Dec 9. PMID 26682756
- [Background] van Leeuwen PJ, Emmett L, Ho B, Delprado W, Ting F, Nguyen Q, Stricker PD. Prospective evaluation of 68Gallium-prostate-specific membrane antigen positron emission tomography/computed tomography for preoperative lymph node staging in prostate cancer. BJU Int. 2017 Feb;119(2):209-215. doi: 10.1111/bju.13540. Epub 2016 Jun 18. PMID 27207581
- [Background] Eiber M, Maurer T, Souvatzoglou M, Beer AJ, Ruffani A, Haller B, Graner FP, Kubler H, Haberkorn U, Eisenhut M, Wester HJ, Gschwend JE, Schwaiger M. Evaluation of Hybrid (6)(8)Ga-PSMA Ligand PET/CT in 248 Patients with Biochemical Recurrence After Radical Prostatectomy. J Nucl Med. 2015 May;56(5):668-74. doi: 10.2967/jnumed.115.154153. Epub 2015 Mar 19. PMID 25791990
- [Background] Afshar-Oromieh A, Avtzi E, Giesel FL, Holland-Letz T, Linhart HG, Eder M, Eisenhut M, Boxler S, Hadaschik BA, Kratochwil C, Weichert W, Kopka K, Debus J, Haberkorn U. The diagnostic value of PET/CT imaging with the (68)Ga-labelled PSMA ligand HBED-CC in the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2015 Feb;42(2):197-209. doi: 10.1007/s00259-014-2949-6. Epub 2014 Nov 20. PMID 25411132
- [Background] Green MA, Eitel JA, Fletcher JW, Mathias CJ, Tann MA, Gardner T, Koch MO, Territo W, Polson H, Hutchins GD. Estimation of radiation dosimetry for 68Ga-HBED-CC (PSMA-11) in patients with suspected recurrence of prostate cancer. Nucl Med Biol. 2017 Mar;46:32-35. doi: 10.1016/j.nucmedbio.2016.11.002. Epub 2016 Nov 4. PMID 28012435

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 68Ga PSMA PET Scan
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 23
Age, Continuous [Median (Full Range); unit: years] | 69 [56 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Ga 68-labeled PSMA-11 Positron Emission Tomography/Computed Tomography (PET/CT) for the Detection on a Per Patient Basis
Description: Sensitivity will be determined on a per-subject basis of 68Ga PSMA PET scan for detection of tumor sites, confirming against imaging, clinical follow-up, and histopathology when available.
Time Frame: Up to 12 months after 68Ga PSMA PET scan
Population: 21 of the 30 subjects had a positive PET/CT scan. 9 of the 21 positive PET/CT scan had enough information to evaluate the results.
Measure: Number; unit: proportion of participants
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 9
proportion of participants | 1.0

2. Secondary Outcome: Positive Predictive Value (PPV) of Ga 68-labeled PSMA-11 Positron Emission Tomography/Computed Tomography (PET/CT) for the Detection of Tumor Location on a Per Patient Basis
Description: Positive predictive value will be determined on a per-subject basis of 68Ga PSMA PET scan for detection of tumor sites, confirming against imaging, clinical follow-up, and histopathology when available.
Time Frame: Up to 12 months after 68Ga PSMA PET scan
Population: as for outcome 1
Measure: Number; unit: proportion of true positives
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 9
proportion of true positives | 1.0

3. Secondary Outcome: Positive Predictive Value (PPV) of Ga 68-labeled PSMA-11 Positron Emission Tomography/Computed Tomography (PET/CT) for the Detection of Prostate Bed Lesions on a Per Patient Basis
Description: as for outcome 2
Time Frame: Up to 12 months after 68Ga PSMA PET scan
Population: 21 of the 30 subjects had a positive PET/CT scan. Five of the 21 positive PET/CT scan had prostate bed lesions, however, only 1 subject had histopathology or Conventional Imaging to confirm positivity.
Measure: Number; unit: proportion of true positives
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 1.0
proportion of true positives | 1.0

4. Secondary Outcome: Positive Predictive Value (PPV) of Ga 68-labeled PSMA-11 Positron Emission Tomography/Computed Tomography (PET/CT) for the Detection of Regional Pelvic Nodal Metastases on a Per Patient Basis
Description: as for outcome 2
Time Frame: Up to 12 months after 68Ga PSMA PET scan
Population: 21 of the 30 subjects had a positive PET/CT scan. Fifteen of the 21 positive PET/CT scan had regional pelvic nodal metastases, however, only 7 subjects had histopathology or Conventional Imaging to confirm positivity.
Measure: Number; unit: proportion of true positives
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 7
proportion of true positives | 1.0

5. Secondary Outcome: Positive Predictive Value (PPV) of Ga 68-labeled PSMA-11 Positron Emission Tomography/Computed Tomography (PET/CT) for the Detection of Extra-pelvic/Visceral Nodal Metastases on a Per Patient Basis
Description: as for outcome 2
Time Frame: Up to 12 months after 68Ga PSMA PET scan
Population: 21 of the 30 subjects had a positive PET/CT scan. 0 of the 21 positive PET/CT scan had detected Extra-pelvic/Visceral Nodal Metastases
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 0

6. Secondary Outcome: Positive Predictive Value (PPV) of Ga 68-labeled PSMA-11 Positron Emission Tomography/Computed Tomography (PET/CT) for the Detection of Osseous Metastases on a Per Patient Basis
Description: as for outcome 2
Time Frame: Up to 12 months after 68Ga PSMA PET scan
Population: 21 of the 30 subjects had a positive PET/CT scan. Six of the 21 positive PET/CT scan had osseous metastases, however, only 2 subject had histopathology or Conventional Imaging to confirm positivity.
Measure: Number; unit: proportion of true positives
Arm/Group | 68Ga PSMA PET Scan
Number analyzed (Participants) | 2
proportion of true positives | 1.0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | 68Ga PSMA PET Scan
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03389451/Prot_SAP_000.pdf